CLINICAL TRIAL: NCT00293631
Title: A Randomized, Parallel-Group, Double-Blind, Single-Dose Study Evaluating the Efficacy and Safety of Intravenous Lornoxicam (8 mg and 16 mg) Compared to Intravenous Placebo and Ketorolac 30 mg in Management of Acute Postoperative Pain Following Orthopedic Surgery (Bunionectomy).
Brief Title: Study of Lornoxicam or Ketorolac or Placebo for Post-Operative Pain After Bunionectomy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: POZEN (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LNP-202
Record Dates: First submitted 2006-02-15; First posted 2006-02-17 (Estimated); Last update posted 2012-12-03 (Estimated); Status verified 2012-11

CONDITIONS: Bunionectomy; Orthopedic Surgery
MeSH Terms: interventions — lornoxicam; Ketorolac

INTERVENTIONS:
Drug: Lornoxicam 8 mg
Drug: Lornoxicam 16 mg
Drug: Ketorolac 30 mg
Drug: Placebo

SUMMARY:
To determine whether a single dose of intravenous lornoxicam is superior to intravenous placebo for management of post-operative pain in patients who have surgical removal of a bunion on the lower extremity. One-fourth of patients in this study will receive a single dose of intravenous ketorolac for management of pain and one-fourth of patients in this study will receive a single dose of an intravenous placebo.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who are scheduled for a primary unilateral first metatarsal bunionectomy under local anesthetic.
* Subjects have no contraindications to this surgery and have no allergies to the study medications or similar medications.
* Subjects are in generally good health with no uncontrolled chronic illnesses or diseases.

Exclusion Criteria:

* Subjects who are pregnant.
* Subjects who have significant obesity.
* Subjects with medically significant heart, liver, kidney, lung or endocrine disease.
* Subjects with active viral disease, i.e. hepatitis, HIV.

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 2005-11; Primary Completion 2006-03 (Actual); Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
The analgesic efficacy (TOTPAR) over 0-12 hours measured on a 100 point Visual Analog Scale (VAS) of a single intravenous dose of lornoxicam (8 mg or 16 mg) compared to placebo in the treatment of post-orthopedic surgery (bunionectomy)
To evaluate the safety and tolerability of lornoxicam administered to subjects with post-bunionectomy surgery pain.

SECONDARY OUTCOMES:
To determine the time to onset of analgesic effect and peak analgesic effect of lornoxicam (8 mg and 16 mg) compared to placebo.

CONTACTS AND LOCATIONS:
Overall Officials: Michael P. DeMicco, MD, Principal Investigator — Advanced Clinical Research Institute
Locations (1):
- Advanced Clinical Research Institute, Anaheim, California, United States